CLINICAL TRIAL: NCT03568760
Title: Finding the Right Words in Neurogenic Communication Disorders: Naming of Objects and Actions, Communicative Strategies in Conversation and Effects of Training
Brief Title: Finding the Right Words in Neurogenic Communication Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-01275
Record Dates: First submitted 2018-05-21; First posted 2018-06-26 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Anomia; Stroke; Aphasia; Parkinson Disease; Multiple Sclerosis
Keywords: Anomia
MeSH Terms: conditions — Anomia; Stroke; Aphasia; Parkinson Disease; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The results are assessed by independent assessors blinded to when the data is obtained and from which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFA treatment (Experimental): Semantic feature analysis
  Interventions: Behavioral: Semantic feature analysis
- Comprehension training (Placebo Comparator): Comprehension training
  Interventions: Behavioral: Comprehension training

INTERVENTIONS:
Behavioral: Semantic feature analysis — Confrontation naming training and training in doing circumlocutions
  Arms: SFA treatment
Behavioral: Comprehension training — Reading and hearing comprehension
  Arms: Comprehension training

SUMMARY:
Every year thousands of persons suffer from brain damage resulting in anomia, that is, word finding difficulties affecting their ability to talk to other people. Anomia may be a result of stroke or of progressive neurological diseases such as Parkinson's disease or multiple sclerosis (MS). Word retrieval is dependent on a complex system of different neural networks and to name objects and activities can be affected to different degrees. The present project explores different aspects of naming ability in altogether 90 persons that has anomia related to stroke or to Parkinson's disease or MS. Furthermore, the communicative strategies and resources used by conversation partners in everyday conversational interaction and in care situations, affected by anomia are studied. Finally, the project includes a study of the effectiveness of a word finding training program based on stimulation of semantic and phonological networks in the brain, involved in the production of words. There is a lack of research on effects on communication from anomia in Parkinson's disease and MS and there is no research on anomia that investigates both object and action naming using a material adapted to the Swedish language. In the project quantitative and qualitative methods are used to explore and describe how persons with different neurogenic communication disorders can use different resources and communicative strategies to express themselves.

DETAILED DESCRIPTION:
Project out line

The main project consists of:

1. A descriptive study of the occurrence and type of naming difficulties in people with stroke, Parkinson's disease or Multiple sclerosis (MS) where quantitative data is compared at group level, (study 1).
2. A descriptive study in which word search strategies are investigated with both quantitative and qualitative methods (study 2).
3. A series of three intervention studies examining the effect of treatment of anomia (studies 3-5).

Study 1: The relation between type of injury and ability to name objects and actions and complex semantic-pragmatic word fluency

Participants The project includes a total of 90 people with anomia: 50 subjects with anomia after stroke, 20 individuals with Parkinson's disease and 20 individuals with MS are recruited are recruited through patient associations and health care facilities in Västra Götaland and included consecutively.

In the study confrontation naming ability, and word fluency is explored. In addition, the type of naming difficulties and consequences of anomia in everyday communication are examined with a questionnaire and communication analysis.

1) Confrontation naming ability is examined with a material consisting of 42 images representing 21 nouns and 21 verbs. The selection of images comes from The Object & Action Naming Battery and is adapted to Swedish linguistic and cultural conditions. The images consist of simple black and white drawings. There is a 20-second time limit for response for each image. In addition to scoring, an analysis and categorization of the response according to the coding scheme is performed; 2) Word fluency is examined with semantic (animals and activities) and phonological (F, A and S) word fluency tests where the participant will produce as many words as possible for each category during one minute. The results are compared with reference data for healthy participants and the use of strategies is analyzed by calculating cluster size and number of switches between different categories; a more complex semantic-pragmatic word fluency task is also administrated.

Participants' experience of their communication skills in everyday life and quality of life is gathered in a questionnaire with image support: The Communication Outcome After Stroke (COAST) scale. COAST consists of 20 questions where participants estimate themselves on a 5-degree likert scale. Stroke and Aphasia Quality of Life Scale (SAQOL-39) and Communicative Participation Item Bank (CPIB) are also administrated as well as a formalized interview.

Study 2: Word search strategies in naming difficulties in people with different types of neurogenic communication disorders

Participants In this descriptive study fifteen participants with Parkinson's disease and fifteen participants with MS are included.

Material and methods Word search strategies in ten-twenty minutes of naturally occurring conversations are assessed through communication analysis. Sequences where participants are involved in repair due to difficulties to express themselves are analyzed with the qualitative method Conversation Analysis in combination med Aktivity based communication analysis.

Studies 3-4: Training with semantic feature analysis to improve naming

Participants Six participants with MS and six participants with Parkinson's disease and 40 participants with anomia due to stroke will be included.

Intervention Participants receive training in semantic feature analysis (SFA) for naming of objects and activities. The training is administered by presenting an image representing either an object or an activity are presented to the participant. The participant is encouraged to try to produce the target word as well as a number of words semantically related to the target word. The related words are listed in a certain order and describe different semantic aspects of the target word. The participants get to choose a number of words which they want to practice.

The participants receive training at 20 occasions, three times a week. The training is delivered during one hour each session in individual training for the participants with MS and in a group setting for two hours, including 30 minutes pause for participants with stroke

Study 3-4 - training anomia due to Parkinson's disease and MS Since semantic feature analysis has not previously been used as treatment for people with Parkinson's disease or MS, the effect is evaluated in using time series design with multiple baselines. Three-five baseline measures of the dependent variable is collected before start of training and then every fourth training session.

Study 5 - training anomia due to stroke In study 5 the effect of intervention for participants with anomia due to stroke is assessed in a randomized group study with a control group. The control group receives training in comprehension. The groups are matched in terms of age, severity of anomia time since onset and level of education. Before and after the intervention, as well as at a twelve week follow up, the effects are assessed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjective experience of word finding difficulties
* Diagnosed left hemisphere stroke or Parkinson's disease or MS
* With correction, sufficient hearing and vision to be able to participate in the assessment
* Participants with stroke at least six months post-onset and documented location of injury.

Exclusion Criteria:

* Mother tongue other than Swedish
* Moderately or severely impaired comprehension
* Other neurological injury or disease
* Moderate-severe apraxia of speech or dysarthria
* Fatigue or impaired attention deficit which prevents participating in intensive training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Naming ability in the Object & Action Naming Battery | At baseline before start of intervention and after 21 days, at completion the intervention program
  A measure of change in ability to name forty pictures consisting of simple black and white drawings. There is a 20-second time limit for response for each picture. Number of correct objects and activities will be calculated separately (range 0-20) as well as summarized (range 0-40)

SECONDARY OUTCOMES:
Sustained change in naming ability in the Object & Action Naming Battery | At a twelve week follow up after the completion of the intervention
  A measure of change in ability to name forty pictures consisting of simple black and white drawings. There is a 20-second time limit for response for each picture. Number of correct objects and activities will be calculated separately (range 0-20) as well as summarized (range 0-40)
Naming of 20 individually chosen training words | At baseline before start of intervention and after 21 days, at completion the intervention program
  A measure of change in ability to name objects and action words participants have chosen to practice
Sustained change in naming of 20 individually chosen training words | At a twelve week follow up after the completion of the intervention
  A measure of change in ability to name objects and action words participants have chosen to practice
The Communication Outcome After Stroke (COAST) scale | At baseline before start of intervention and after 21 days, at completion the intervention program
  A measure of change in participants perception of the communicative ability from baseline to after intervention. COAST comprises 20 items where participants rates themselves on a 5-graded likert scale. The scale is running from 1) "couldn't do it at all, through 2) "with a lot of difficulty", 3) "with some difficulty", 4) "quite well" to 5) "very well". The scoring of each item will be summarized and averaged (total range 0-5) and a higher score indicates perceptions of better communicative ability.
Sustained change in the Communication Outcome After Stroke (COAST) scale | At a twelve week follow up after the completion of the intervention
  A measure of change in participants perception of the communicative ability twelve weeks after intervention is completed. COAST comprises 20 items where participants rates themselves on a 5-graded likert scale. The scale is running from The scale is running from 1) "couldn't do it at all, through 2) "with a lot of difficulty", 3) "with some difficulty", 4) "quite well" to 5) "very well". The scoring of each item will be summarized and averaged (total range 0-5) and a higher score indicates perceptions of better communicative ability.
The Stroke Aphasia Quality of Life (SAQOL-39) | At baseline before start of intervention and after 21 days, at completion the intervention program
  A measure of change after intervention in participant reported health related quality of life in a questionnaire with 39 items where participants evaluate of their everyday functioning in three domains: physical, psychosocial and communication. Scores range from 1 to 5 in each sub domain and are averaged; higher scores indicate better quality of life. Scoring in each domain will be summarized and averaged and presented separately as well as in a compound averaged score (range 1-5).
Sustained change in the Stroke Aphasia Quality of Life (SAQOL-39) | At a follow up twelve weeks after completion of intervention
  A measure of change 12 weeks after intervention is completed in participant reported health related quality of life in a questionnaire with 39 items where participants evaluate of their everyday functioning in three domains: physical, psychosocial and communication. Scores range from 1 to 5 in each sub domain and are averaged; higher scores indicate better quality of life. Scoring in each domain will be summarized and averaged and presented separately as well as in a compound averaged score (range 1-5).
The Communicative Participation Item Bank (CPIB) | At baseline before start of intervention and after 21 days, at completion the intervention program
  A measure of change from baseline to after intervention in participants' perceptions of their communicative participation in everyday life activities. A short form of the item bank with ten items are used - participants rates their perception of degree of participation on a four-graded scale where higher scores indicate higher degree of participation. The scale runs from 0) "very much", through 1) "quite a bit", 2) "a little", to 3) "not at all". The scoring of each item will be summarized into a total score (range 0-30).
Sustained change in the Communicative Participation Item Bank (CPIB) | At a 12 week follow up after the completion of the intervention
  A measure of change 12 weeks after the completion of the intervention in participants' perceptions of their communicative participation in everyday life activities. A short form of the item bank with ten items are used - participants rates their perception of degree of participation on a four-graded scale where higher scores indicate higher degree of participation. The scale runs from 0) "very much", through 1) "quite a bit", 2) "a little", to 3) "not at all". The scoring of each item will be summarized into a total score (range 0-30).
Retelling of events in video clips | At baseline before start of intervention and after 21 days, at completion the intervention program
  A measure of change in ability to retell and describe events from baseline to after intervention is completed.The participants view short video clips with a character involved with different activities including objects and are asked to retell what happened every tenth second.
Sustained change in retelling of events in video clips | At a 12 week follow up after the completion of the intervention
  A measure of change in ability to retell and describe events from after the completion of intervention to a 12 weeks follow up. The participants view short video clips with a character involved with different activities including objects and are asked to retell what happened every tenth second.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta Saldert, Principal Investigator — Inst of Neurosci & Physiology, Speech & Language Pathology Unit University of Gothenburg
Locations (1):
- University of Gothenburg, Gothenburg, Västra Göraland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tallberg IM, Ivachova E, Jones Tinghag K, Ostberg P. Swedish norms for word fluency tests: FAS, animals and verbs. Scand J Psychol. 2008 Oct;49(5):479-85. doi: 10.1111/j.1467-9450.2008.00653.x. Epub 2008 Apr 29. PMID 18452499
- [Background] Long A, Hesketh A, Paszek G, Booth M, Bowen A. Development of a reliable self-report outcome measure for pragmatic trials of communication therapy following stroke: the Communication Outcome after Stroke (COAST) scale. Clin Rehabil. 2008 Dec;22(12):1083-94. doi: 10.1177/0269215508090091. PMID 19052247
- [Background] Baylor C, Yorkston K, Eadie T, Kim J, Chung H, Amtmann D. The Communicative Participation Item Bank (CPIB): item bank calibration and development of a disorder-generic short form. J Speech Lang Hear Res. 2013 Aug;56(4):1190-208. doi: 10.1044/1092-4388(2012/12-0140). Epub 2013 Jul 1. PMID 23816661
- [Background] Hilari K, Lamping DL, Smith SC, Northcott S, Lamb A, Marshall J. Psychometric properties of the Stroke and Aphasia Quality of Life Scale (SAQOL-39) in a generic stroke population. Clin Rehabil. 2009 Jun;23(6):544-57. doi: 10.1177/0269215508101729. Epub 2009 May 15. PMID 19447841